CLINICAL TRIAL: NCT04029584
Title: The Effects of Single Dose Rifampin on Pharmacokinetics of Fluvastatin in Uninduced and Hepatically Induced Healthy Volunteers
Brief Title: Drug-Drug Interaction Between Rifampin and Fluvastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18-27008
Record Dates: First submitted 2019-07-16; First posted 2019-07-23 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Drug-drug Interaction
Keywords: drug-drug interaction; statin; rifampin
MeSH Terms: interventions — Rifampin; Fluvastatin

STUDY DESIGN:
Intervention Model Description: This study is a two arm, randomized, open label, crossover, clinical trial. Arm 1 will be conducted in normal healthy volunteers; Arm 2 will be conducted in hepatically induced (by oral rifampin) healthy volunteers.
Masking Description: No masking will be employed because it is very difficult to mask the effects of rifampin (range discoloration) on subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fluvastatin Alone First, Then Fluvastatin +IV Rifampin 600 mg (Experimental): The effect of rifampin on the pharmacokinetics of fluvastatin will be studied in healthy volunteers with or without hepatic induction in a randomized, unblinded, crossover clinical trial.
  For uninduced periods, subjects will be randomized to receive one oral dose of fluvastatin (Lescol®) 20mg capsule first. Separated by one day of washout, they then receive one oral dose of fluvastatin (Lescol®) 20mg capsule immediately following a 30-min intravenous infusion of rifampin 600mg in 10ml Normal Saline.
  Before starting hepatic induced period, subjects will have a washout for greater than one week.
  To induce hepatic enzyme and transporter, Subjects will be pretreated with 5 days with 600mg oral rifampin. Subjects will be then randomized first to receive a single dose of fluvastatin 20mg. Separated by one day of washout, subject will then receive one oral dose of fluvastatin 20mg immediately after a 30-min IV infusion of rifampin 600mg.
  Interventions: Drug: rifampin IV; Drug: Rifadin 300Mg Capsule; Drug: Fluvastatin 20 MG
- Fluvastatin +IV Rifampin 600 mg First, Then Fluvastatin Alone (Experimental): The effect of rifampin on the disposition of fluvastatin will be studied in healthy volunteers with or without hepatic induction in a randomized, unblinded, crossover clinical trial.
  For uninduced periods, subjects will be randomized to first receive one oral dose of fluvastatin (Lescol®) 20mg capsule immediately following a 30-min intravenous infusion of rifampin 600mg in 10ml Normal Saline.Separated by one day of washout, subjects will be then receive a single dose of fluvastatin (Lescol®) 20mg capsule.
  Before starting induction periods, subjects will have a washout greater than one week.
  To induce hepatic enzyme and transporter, subjects will be pretreated with 5 days with 600mg oral rifampin. subjects will be randomized to receive first one oral dose of fluvastatin 20mg immediately after a 30-min IV infusion of rifampin 600mg. Separated by one day of washout, subject will then receive one oral dose of fluvastatin 20mg.
  Interventions: Drug: rifampin IV; Drug: Rifadin 300Mg Capsule; Drug: Fluvastatin 20 MG

INTERVENTIONS:
Drug: rifampin IV — A 30-min intravenous infusion of rifampin 600mg in 10ml Normal Saline will be used to inhibit hepatic OATP1B1 transporters.
Drug: Rifadin 300Mg Capsule — Rifadin 600mg by mouth as two 300mg rifadin capsules
Drug: Fluvastatin 20 MG — one oral dose of fluvastatin (Lescol ) 20mg capsule

SUMMARY:
The effect of organic anion transporting polypeptide 1B1 (OATP1B1) transporter inhibition at clinical doses of fluvastatin, a biopharmaceutics drug disposition classification system (BDDCS) class 1 drug, has not been studied to date. A single dose of IV rifampin can be used as model OATP1B1 inhibitor to evaluate the significance of OATP1B1 transporter effects on fluvastatin disposition. A preinduction regimen of oral rifampin followed by a single IV infusion of rifampin can be used to evaluate the combined effects of enzyme induction and OATP1B1 transporter inhibition on fluvastatin disposition. A two arm, randomized, open label, crossover clinical study in healthy, volunteers will be conducted to evaluate the effects of IV rifampin on fluvastatin disposition in both hepatically induced and uninduced subjects.

DETAILED DESCRIPTION:
The effect of rifampin on the pharmacokinetics of fluvastatin will be studied in healthy volunteers in a two arms, two-period, randomized, unblinded, crossover clinical trial. In the first arm, subjects will be randomized to one of two treatment groups:

(i)fluvastatin (Lescol®) 20mg capsule (ii) one oral dose of fluvastatin (Lescol®) 20mg capsule immediately following a 30-min intravenous infusion of rifampin 600mg in 10ml Normal Saline.

In the second arms, patients will be pretreated with 600mg oral rifampin (two 300mg rifadin capsule) once daily to induce hepatic enzymes (and transporters) for 5 years. Subjects will be randomized to one of two treatment groups:

(i) one oral dose of fluvastatin (Lescol®) 20mg capsule (ii) one oral dose of fluvastatin (Lescol®) 20mg capsule immediately following a 30-min intravenous infusion of rifampin 600mg in 10ml Normal Saline

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, ages 18-65 years old, with no current medical conditions or active diagnoses as determined by the study doctor based on history, physical exam, and laboratory evaluations.
2. Subjects who take no other medications two weeks prior to the study and during the time course of the study including prescription medications, over-the-counter medications, dietary supplements, or drugs of abuse.
3. Subjects able to maintain adequate birth control during the study independent of hormonal contraceptives (including hormonal intrauterine devices (IUDs)). Adequate methods of contraception include use of condoms and copper IUDs.
4. Subjects able to abstain from grapefruit, grapefruit juice, oranges, orange juice, caffeinated beverages and/or alcoholic beverages from 7am the day before the study to completion of that study day.
5. Participants determined to have normal liver and kidney function as measured at baseline ( alanine aminotransferase (ALT): ≤ 2x upper level of normal (ULN), aspartate aminotransferase (AST): ≤ 2x ULN, serum creatinine (SCr): ≤ 1.5x ULN, T. Bili: 0.1-1.2mg/dL, Albumin: 3.4 - 4.7 mg/dL).
6. BMI between 18.0 - 30 kg/m2 o Subjects capable of fasting from food and beverages at least 8 hours prior to medication dosing.
7. Be able to read, speak, and understand English.
8. Subjects capable of providing informed consent and completing the requirements of the study.

Exclusion Criteria:

1. Subjects with active medical problems
2. Subjects on chronic prescription or over the counter (OTC) medication that cannot be stopped 2 weeks prior to and during the study.
3. Subjects incapable of multiple blood draws (HCT < 30mg/dL)
4. Subjects with a history of rhabdomyolysis
5. Subjects with a history of drug-related myalgias
6. Subjects with a history or diagnosis of hemorrhagic tendencies or blood dyscrasias
7. Subjects with a history of GI bleed or peptic ulcer disease
8. Subjects who smoke tobacco or have ongoing alcohol or illegal drug use
9. Subjects who are pregnant, lactating, or trying to conceive during the study period
10. Subjects allergic to fluvastatin or rifampin or any known component of the medications
11. Anyone who in the opinion of the study investigators is unable to do the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Benet, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
All study data will be stored and analyzed at University of California San Francisco (UCSF) by the Principal investigator and Key Study personnel. There are no plans of sharing the subjects data with any outside entities.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Flyer on campus and Craiglist
Pre-assignment Details: During the uninduced and induced study interventions there were separate randomization procedures.
Groups:
- Fluvastatin Alone First, Then Fluvastatin +IV Rifampin 600 mg: Subjects received one oral dose of fluvastatin (Lescol®) 20mg capsule.
- Fluvastatin +IV Rifampin 600 mg First, Then Fluvastatin Alone: Subjects received one oral dose of fluvastatin (Lescol®) 20mg capsule immediately following a 30-min intravenous infusion of rifampin 600mg in 10ml Normal Saline.
Period: Uninduced Study 1st Intervention (1 Day)
Arm/Group | Fluvastatin Alone First, Then Fluvastatin +IV Rifampin 600 mg | Fluvastatin +IV Rifampin 600 mg First, Then Fluvastatin Alone
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0
Period: Uninduced Washout (1 Day)
Arm/Group | Fluvastatin Alone First, Then Fluvastatin +IV Rifampin 600 mg | Fluvastatin +IV Rifampin 600 mg First, Then Fluvastatin Alone
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0
Period: Uninduced Study 2nd Intervention (1 Day)
Arm/Group | Fluvastatin Alone First, Then Fluvastatin +IV Rifampin 600 mg | Fluvastatin +IV Rifampin 600 mg First, Then Fluvastatin Alone
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0
Period: Washout Between (>1 Week)
Arm/Group | Fluvastatin Alone First, Then Fluvastatin +IV Rifampin 600 mg | Fluvastatin +IV Rifampin 600 mg First, Then Fluvastatin Alone
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0
Period: Induced Study 1st Intervention (1 Day)
Arm/Group | Fluvastatin Alone First, Then Fluvastatin +IV Rifampin 600 mg | Fluvastatin +IV Rifampin 600 mg First, Then Fluvastatin Alone
Started | 2 | 8
Completed | 2 | 8
Not Completed | 0 | 0
Period: Induced Washout (1 Day)
Arm/Group | Fluvastatin Alone First, Then Fluvastatin +IV Rifampin 600 mg | Fluvastatin +IV Rifampin 600 mg First, Then Fluvastatin Alone
Started | 2 | 8
Completed | 2 | 8
Not Completed | 0 | 0
Period: Induced Study 2nd Intervention (1 Day)
Arm/Group | Fluvastatin Alone First, Then Fluvastatin +IV Rifampin 600 mg | Fluvastatin +IV Rifampin 600 mg First, Then Fluvastatin Alone
Started | 2 | 8
Completed | 2 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy volunteers
Groups:
- All Subjects: Subjects were randomized to one of two treatment groups: 1) a single oral dose of fluvastatin (Lescol®) 20 mg capsule or 2) a single oral dose of fluvastatin (Lescol®) 20 mg capsule immediately following a 30-min intravenous infusion of rifampin 600 mg in 10 mL normal saline.
Arm/Group | All Subjects
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 4
  African American | 2
  Asian | 2
  Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 10
Serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.79 (0.13)

OUTCOME MEASURES:

1. Primary Outcome: AUC
Description: The primary outcome will be fluvastatin Area under the concentration vs time curve (AUC0-12h and AUC0-INF)
Time Frame: AUC will be assessed over a 12 hour study at 0, 0.33, 0.67,1,1.5, 2, 2.5, 3, 4, 6, 9, 12h
Population: healthy volunteer
Measure: Mean (Standard Deviation); unit: ng/mL·h
Groups:
- Fluvastatin Control: healthy volunteer take a single dose fluvastatin
- Fluvastatin and IV Rifampin: Healthy volunteer takes a single IV rifampin prior to oral fluvastatin
- Fluvastatin + Oral Rifampin Induction: Healthy volunteers who take oral rifampin for 5 days prior to oral fluvastatin
- Fluvastatin +Oral Rifampin Induced +IV Rifampin: Healthy takes five days oral rifampin, and then take one oral dose of fluvastatin (Lescol®) 20mg capsule immediately following a 30-min intravenous infusion of rifampin 600mg in 10ml Normal Saline
Arm/Group | Fluvastatin Control | Fluvastatin and IV Rifampin | Fluvastatin + Oral Rifampin Induction | Fluvastatin +Oral Rifampin Induced +IV Rifampin
Number analyzed (Participants) | 10 | 10 | 10 | 10
ng/mL·h
  AUC(0-12) | 242 (83) | 642 (269) | 124 (33.7) | 371 (217)
  AUC(0-INF) | 266 (86) | 679 (274) | 136 (35.9) | 385 (222)

2. Secondary Outcome: Cmax
Description: Secondary outcomes will include fluvastatin maximum plasma concentration (Cmax).
Time Frame: Cmax will be assessed over a 12 hour study period.
Population: healthy volunteers
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fluvastatin Control | Fluvastatin and IV Rifampin | Fluvastatin + Oral Rifampin Induction | Fluvastatin +Oral Rifampin Induced +IV Rifampin
Number analyzed (Participants) | 10 | 10 | 10 | 10
ng/mL | 176 (149) | 447 (342) | 87.8 (37.3) | 379 (446)

3. Secondary Outcome: Tmax
Description: Secondary outcomes will include time to Cmax (Tmax).
Time Frame: Tmax will be assessed over a 12 hour study period.
Population: healthy volunteer
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Fluvastatin Control | Fluvastatin and IV Rifampin | Fluvastatin + Oral Rifampin Induction | Fluvastatin +Oral Rifampin Induced +IV Rifampin
Number analyzed (Participants) | 10 | 10 | 10 | 10
hr | 1.20 (0.62) | 1.17 (0.72) | 1.28 (0.545) | 1.23 (0.960)

ADVERSE EVENTS:
Time Frame: Adverse event was monitored in uninduced arm from study day 1 to day 3. Adverse event was monitored in induced arm from study day -5 to day 3.
Groups:
- Uninduced Healthy Volunteer Fluvastatin Alone: Subjects randomized to receive one oral dose of fluvastatin (Lescol®) 20mg capsule
- Uninduced Healthy Volunteer Fluvastatin and Rifampin: Subjects randomized to receive one oral dose of fluvastatin 20mg immediately after a 30-min IV infusion of rifampin 600mg.
- Hepatic Induced Healthy Volunteer Fluvastatin Alone: Subjects pretreated with 5 days with 600mg oral rifampin for enzyme and transporter induction. Subjects randomized to receive one oral dose of fluvastatin 20mg
- Hepatic Induced Healthy Volunteer Fluvastatin and Rifampin: Subjects pretreated with 5 days with 600mg oral rifampin for enzyme and transporter induction. Subjects randomized to receive one oral dose of fluvastatin 20mg immediately after a 30-min IV infusion of rifampin 600mg.
Arm/Group | Uninduced Healthy Volunteer Fluvastatin Alone | Uninduced Healthy Volunteer Fluvastatin and Rifampin | Hepatic Induced Healthy Volunteer Fluvastatin Alone | Hepatic Induced Healthy Volunteer Fluvastatin and Rifampin
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT04029584/Prot_SAP_001.pdf
  • Informed Consent Form (2018-12-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT04029584/ICF_002.pdf